CLINICAL TRIAL: NCT00500968
Title: Randomized Study Assessing the Effect of Transpapillary Pancreas Duct Stent in Resection of the Pancreatic Tail
Brief Title: Study Assessing the Effect of Transpapillary Pancreas Duct Stent in Resection of the Pancreatic Tail
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Karolinska Institutet (Other)
Responsible Party: Karoliska instuitut, Farshad Frozanpor
Allocation: Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2006/3:3
Record Dates: First submitted 2007-07-12; First posted 2007-07-13 (Estimated); Last update posted 2011-04-07 (Estimated); Status verified 2007-09

CONDITIONS: Pancreas Cancer; Fistula
Keywords: Pancreas; Leakage; Fistula; tail
MeSH Terms: conditions — Pancreatic Neoplasms; Fistula | interventions — Stents; Cholangiopancreatography, Endoscopic Retrograde; Surgical Procedures, Operative

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Stent (Active Comparator)
  Interventions: Procedure: stent
- conventional distal pancreatectomy (Active Comparator)
  Interventions: Procedure: Distal pancreatectomy

INTERVENTIONS:
Procedure: stent — ERCP guided stent insertion before transection of the gland
  Other Names: ERCP
  Arms: Stent
Procedure: Distal pancreatectomy — conventional distal pancreatectomy
  Other Names: surgery
  Arms: conventional distal pancreatectomy

SUMMARY:
Randomized study assessing the effect of transpapillary pancreas duct stent in resection of the pancreatic tail.

DETAILED DESCRIPTION:
Resection of the pancreatic tail is fraught with fistula or leakage of pancreatic enzymes to varying degrees between 13-64%, depending upon which definition one uses. The "downstream" control of the pancreatic duct with the help of a transpapillary stent might minimize the risk for leakage over the transected pancreas surface.

Trial evaluation will be A. The pancreatic bed was drained and postoperatively the fluid was continuously collected and daily analysed for pancreatic amylase and bilirubin. Daily measurement of pancreatic enzyme content in the drain fluid, at least for 5 post operative days or as long as the patient retains the drain. X-Amylase and X-Protein as long as the patient has the external drain.

B. Co-variables measured in the form of: operation time, complications in relation to diagnosis, duration of hospitalization. Patients receiving a pancreas stent are followed in order to evaluate the natural course of the pancreas stent.

ELIGIBILITY:
Inclusion Criteria:

* Inclusion Criteria include all patients planned to undergo resection of the pancreatic body-tail are invited to participate.

Exclusion Criteria:

* The Patients who, at the time of exploration, judged to have a tumour, which is un-resectable.

Min Age: 20 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50 (Actual)
Dates: Start 2006-11; Primary Completion 2011-04 (Actual); Study Completion 2011-04 (Actual)

PRIMARY OUTCOMES:
Drain fluid content analyses | At least 5 postoperative days
  Post-operative daily measurement of X-Amylase,as long as the patient has the external drain and for at least 5 postopertaive days.

SECONDARY OUTCOMES:
Co-variables measured in the form of: operation time, complications in relation to diagnosis, duration of hospitalization and cost. Patients receiving a pancreas stent are followed in order to evaluate the natural course of the pancreas stent | At least 5 postoperative days

CONTACTS AND LOCATIONS:
Overall Officials: Urban Arnelo, Study Director — Karolinksa university hospital; Farshad Frozanpor, Principal Investigator — Karolinksa university hospital; Lars Lundell, Professor, Study Chair — Karolinska Institutet
Locations (1):
- Karolinksa university hospital, Stockholm, Sweden

REFERENCES:
- [Derived] Frozanpor F, Lundell L, Segersvard R, Arnelo U. The effect of prophylactic transpapillary pancreatic stent insertion on clinically significant leak rate following distal pancreatectomy: results of a prospective controlled clinical trial. Ann Surg. 2012 Jun;255(6):1032-6. doi: 10.1097/SLA.0b013e318251610f. PMID 22584629